CLINICAL TRIAL: NCT04916054
Title: Time to Surgery and Survival Outcomes for Patients With Resected Colorectal Carcinoma: Multicenter Study (BIG RENAPE)
Acronym: DELARC
Status: Completed | Type: Observational
Sponsor: Institut Cancerologie de l'Ouest (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: ICO-2021-10
Record Dates: First submitted 2021-06-01; First posted 2021-06-07 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2021-05

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Colorectal cancer (CRC) is diagnosed in one million patients each year worldwide and is the 2nd leading cause of cancer death. Peritoneal metastasis (MP) is seen in 10% of CRC patients and is the metastatic site with the worst prognosis.

Complete cytoreduction surgery (CCS) is the only treatment that allows for prolonged survivals. Five-year overall survival (OS) after CCS ranges from 30% to 60% compared with 0 to 5% with exclusive medical treatment.

Chemotherapy (CT) with fluoropyrimidine and oxaliplatin and/or irinotecan 3 months pre-operatively and 3 months adjuvant is widely used. The benefits of perioperative CT have been demonstrated in another resectable metastatic site, the liver and has become by extension a therapeutic standard in France for CRC MPs. However, the impact of delay in the initiation of surgery and adjuvant or neoadjuvant CT is unknown for CRC MPs.

Several deleterious oncologic effects are related to a long period without treatment between

* Neoadjuvant chemotherapy and surgery:
* Surgery and adjuvant chemotherapy.

Several meta-analyses have demonstrated, for at least 13 different cancers, a continuous association between delays in treatment (CT, radiotherapy, or surgery) and cancer mortality. For CRC, Hanna's meta-analysis showed that for every 4-week delay in adjuvant surgery or CT, the risk of cancer death increased by 6 and 13%, respectively.

These long delays between CT and excisional surgery also decrease survival in patients with liver metastases from colorectal origins and MPs from ovarian origins but this has never been evaluated in patients with MPs from colorectal origins.

Demonstrating an oncologic impact of therapeutic delays would have several strategic practical impacts such as:

* Promoting pre- and post-operative rehabilitation programs to facilitate recovery and reduce time to retreatment.
* To use more easily techniques (protective stoma, multi-stage surgery) limiting the risk of complications and therefore the delays in treatment.
* Propose clinical research protocols aimed at reducing these delays with knowledge of plausible statistical hypotheses.

A therapeutic strategy of shortening the time between each treatment therefore deserves to be evaluated in metastatic forms of colorectal cancer.

The investigators would like to evaluate the hypothesis that shortened time between treatments could have a prognostic impact on recurrence-free survival.

DETAILED DESCRIPTION:
This is a retrospective study including exhaustively all patients operated CC0-CC1 of peritoneal carcinosis between 2007 and 2019 meeting the inclusion criteria:

* Patients from the Institut de cancérologie de l'Ouest and the CHU of Lyon for the study period 2007-2016
* Patients included in the BIG-RENAPE network between 2016 and 2019

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years
2. Histological evidence of peritoneal metastases
3. Primary colorectal cancer
4. Surgical cytoreduction CC0 or CC1

Exclusion Criteria:

1. Patient who has not received at least 3 courses of pre and/or post cytoreduction chemotherapy
2. Primitive appendicitis
3. Unknown primitive
4. Patient with incomplete CC2 and/or palliative surgery
5. Patient opposed to the use of their data for research.
6. Isolated local pelvic recurrence.
7. Extraperitoneal metastases not resected or destroyed before or during cytoreduction.
8. Patient opposed to the use of his/her data for research purposes

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patient with a surgery for peritoneal carcinosis of colorectal origin between 2007 and 2019
  * Patients from the Institut de cancérologie de l'Ouest and the CHU of Lyon for the study period 2007-2016
  * Patients included in the BIG-RENAPE network between 2016 and 2019
Sampling Method: Non-Probability Sample
Enrollment: 227 (Actual)
Dates: Start 2021-06-04 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-03-10 (Actual)

PRIMARY OUTCOMES:
to determine whether the time between each anti-tumor therapy has a prognostic impact on recurrence-free survival | 2 years
  recurrence-free survival

SECONDARY OUTCOMES:
To evaluate the impact on overall survival | 2 years
  overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric DUMONT, MD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (2):
- France (2):
  - CHU LYON, Lyon
  - Institut de Cancerologie de L'Ouest, Saint-Herblain

IPD SHARING:
Plan to Share IPD: No